CLINICAL TRIAL: NCT03545308
Title: Pharmacokinetics of Rocuronium (1 mg/kg) for Deep Block : a Prospective Observational Study
Brief Title: Pharmacokinetics of Rocuronium for Deep Block (DeepRocu)
Acronym: DeepRocu
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Principal Investigator, Philippe Cuvillon, Clinical Professor (PhD), Centre Hospitalier Universitaire de Nīmes
Other Study IDs: 2016-01-01
Record Dates: First submitted 2017-12-29; First posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-06

CONDITIONS: Neuromuscular Blockade
Keywords: Neuromuscular; Deep Anesthesia; Rocuronium
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Rocuronium — Dose: 1 mg/kg

SUMMARY:
Rocuronium is a non-depolarising neuromuscular blocking agent. The compound has a rapid onset and an intermediate duration of action.

The rapid onset is of importance in patients at risk for pulmonary aspiration, for elective induction of anesthesia. Clinical studies simulating rapid sequence induction in elective patients indicate that rocuronium 0.9 mg kg-1 may be suitable for crash intubation.Also, rocuronium may be an alternative to succinylcholine for rapid sequence induction when high dose is injected (3x Effective Dose 95 %= 1mg/kg). But, pharmacokinetic of rocuronium at 1 mg/kg is not well establish.

The investigator investigate the onset and recovery of a single dose rocuronium (1 mg/kg) in consecutive patients (>100) using adductor muscle monitoring (Train of Four and Post Tetanic Count)

DETAILED DESCRIPTION:
In this study, pharmacokinetic of rocuronium at 1 mg/kg will be evaluated at each point of Train of Four Response (TOF) and Post Tetanic Count (when TOF=0) troughout the period of anesthesia and surgery.

Time 0 is the time of rocuronium injection, Time 1 is the time when post tetanic count is > 5-7 and TOF=0, Time 3 when TOF >0 response, Time 4 when 4 reponses of the TOF and Time 5 when TOF > 90 %

ELIGIBILITY:
Inclusion Criteria:

* elective or emergency surgery under general anesthesia with deep block
* approval
* adult

Exclusion Criteria:

* contra indication to neuromuscular blockade (allergy, myopathy, hyperkaliemia)
* refusal
* < 18 years olds
* Body mass index > 50
* neuropathy
* regional anesthesia

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for surgery under general anesthesia with the need of deep neuromuscular block for surgery
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Onset | 3 hour
  The elapsed time (in minute) between Time 0 (injection of rocuronium) to T1 (PTC > 5-7)

SECONDARY OUTCOMES:
intubation | 1 hour
  time for intubation
Post Tetanic Count recovery | 3 hours
  Times between Post Tetanic Count = 0 to 20 (Time 3)
Recovery Train of Four | 6 hours
  Times between T0 to train of four= 4 (Time 4)
Antagonization | 6 hours
  Evaluation of recovery with sugammadex or prostigmine

CONTACTS AND LOCATIONS:
Overall Officials: jean-yves lefrant, MD,PhD, Study Chair — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU Nimes, Nîmes, Gard, France

IPD SHARING:
Plan to Share IPD: No